CLINICAL TRIAL: NCT02245451
Title: A Single-centre, Open-label Study of Multiple Doses of Tipranavir 500 mg and Ritonavir 200 mg (Twice Daily) on the Pharmacokinetic Characteristics of Methadone Administered as a Single Dose in Healthy Volunteers
Brief Title: Study of Tipranavir and Ritonavir on the Pharmacokinetic Characteristics of Methadone Administered in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.26
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Methadone

ARMS (1):
- TPV/r with methadone (Experimental)
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Methadone

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Methadone

SUMMARY:
The primary objective of this study is to characterise the effects of tipranavir 500 mg and ritonavir 200 mg (TPV/r; given twice daily) at steady-state on the pharmacokinetics of methadone administered as a single dose in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers aged at least 18 to 60 years.
* Clinically normal medical history.
* Clinically normal findings on physical examination.
* Clinically normal laboratory values.
* A Body Mass Index >18.5 and <30 kg/m2.
* Able to swallow large capsules without difficulty.
* Capable of comprehending and communicating effectively with the investigator and staff and of providing written informed consent in accordance with ethics committee and regulatory guidelines.
* Willing to stay in the study centre for the duration of the study.
* Willing to abstain from ingesting substances during the study which may alter plasma study drug levels by interaction with the cytochrome P450 system.
* Willing to abstain from alcohol for 48 hours prior to Visit 1 and for the duration of the study. In addition, Cabernet Sauvignon must not have been ingested within 15 days prior to Visit 1.
* Willing to abstain from ingesting grapefruit and grapefruit juice for 15 days before Visit 1 and for the duration of the study.
* Willing to abstain from ingesting Seville oranges, strawberries or strawberry extract, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) for 72 hours before the pharmacokinetic sampling days.
* Willing to abstain from use of tobacco products for the duration of the study.
* Urine drug screen negative for illegal non-prescription drugs.
* Negative HIV serology.
* Negative for Hepatitis B surface antigen and Hepatitis C

Exclusion Criteria:

* Any clinically significant disease. (A significant disease was defined as a disease which in the opinion of the investigator may either have put the subject at risk because of participation in the study or a disease which may have influenced the results of the study or the subject's ability to participate in the study.)
* Clinically significant abnormal baseline haematology, blood chemistry or urinalysis findings.
* Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), cholesterol, triglyceride or glucose greater than the upper limit of normal at Visit 1.
* Treatment with prohibited medications in the thirty days before the study or during the study or ingestion of drugs of abuse.
* Treatment with any investigational drug within 90 days of the first dose of study medication.
* Inability to adhere to the requirements of the protocol (including active substance abuse) as assessed by the investigator.
* Prior tipranavir use.
* Ingestion of any known enzyme altering drug (such as phenothiazines, cimetidine, barbiturates, ketoconazole, fluconazole, clarithromycin, rifampin, steroids, and herbal medications) for thirty days prior to Visit 1.
* Ingestion of grapefruit, grapefruit juice, and Cabernet Sauvignon within fifteen days prior to Visit 1.
* Ingestion of Seville oranges, strawberries or strawberry extract, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc) within 72 hours of pharmacokinetics sampling days.
* Treatment with prescription medicines within thirty days prior to Visit 1.
* History of gastrointestinal, hepatic, or renal disorders within 60 days prior to Visit 1.
* Any history of alcohol or drug abuse.
* Current use of cigarettes defined as greater than 10 cigarettes per day or rolling/pipe tobacco equivalent.
* Blood or plasma donations within 90 days prior to Visit 1
* Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >100 beats/min.
* Subjects with a history of any illness or allergy that, in the opinion of the investigator, might have confounded the results of the study or posed additional risk in administering tipranavir, ritonavir or methadone to the subject.
* Subjects who had an acute illness within two weeks prior to Visit 1.
* Subjects who were currently taking any over-the-counter drug within fourteen days prior to Visit 1 or who were currently taking any prescription drug.
* Hypersensitivity to tipranavir, ritonavir, or methadone.
* Female subjects who are of reproductive potential and who were pregnant, breastfeeding, had a positive serum B-HCG at Visit 1 or 2, had not been using a barrier contraceptive method for at least three months prior to Study Day 1 or were not willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam) during the study and for thirty days after completion or termination of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-01; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve for 0 to 24 hours (AUC0-24h) of methadone | up to 24 hours after drug administration
Maximum concentration (Cmax) | up to 24 hours after drug administration
Concentration at 6 hours (C6h) of methadone | 6 hours after drug administration
Area under the concentration-time curve for 0 to 12 hours (AUC0-12h) of tipranavir and ritonavir | up to 12 hours after drug administration
concentration at 12 hours (C12h) of tipranavir and ritonavir | 12 hours after drug administration

SECONDARY OUTCOMES:
mean residence time (MRT) | up to 24 hours after drug administration
apparent terminal half-life (t½) | up to 24 hours after drug administration
time to maximum concentration (Tmax) | up to 24 hours after drug administration
oral clearance (CL/F) | up to 24 hours after drug administration
apparent volume of distribution during the terminal elimination phase divided by the bioavailability factor (Vz/F) | up to 24 hours after drug administration
Number of patients with abnormal findings in physical examination | Up to day 17 after first drug administration
Number of patients with clinically significant changes in vital signs | Up to day 17 after first drug administration
Number of patients with abnormal changes in clinical laboratory parameters | Up to day 17 after first drug administration
Number of participants with adverse events | Up to day 17 after first drug administration